CLINICAL TRIAL: NCT07009145
Title: An Exploratory Study of Iparomlimab and Tuvonralimab (QL1706) in Combination With Bevacizumab for the Treatment of Unresectable or Metastatic MSI-H/dMMR Colorectal Cancer
Brief Title: QL1706 Plus Bevacizumab for Unresectable or Metastatic MSI-H/dMMR CRC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Collaborators: Linyi Tumour Hospital (Other); Shandong Provincial Hospital (Other Government); Qingdao Central Hospital (Other)
Responsible Party: Principal Investigator, Jun Wang, Associate Director, Department of Oncology, Qianfoshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2025(092)
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Unresectable Colorectal Cancer; Metastatic Colorectal Cancer (CRC); MSI-H/dMMR Colorectal Cancer
Keywords: QL1706; CRC; MSI-H/dMMR
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 + Bevacizumab (Experimental)
  Interventions: Drug: QL1706; Drug: Bevacizumab

INTERVENTIONS:
Drug: QL1706 — QL1706 (Iparomlimab and Tuvonralimab) is administered at a dose of 5 mg/kg via intravenous infusion on Day 1 of each 3-week cycle (Q3W).
Drug: Bevacizumab — Bevacizumab is administered at a dose of 7.5 mg/kg every 3 weeks (Q3W) via intravenous (iv) infusion.

SUMMARY:
This is a single-arm, multi-center, exploratory study evaluating the efficacy and safety of iparomlimab and tuvonralimab (QL1706) in combination with bevacizumab for the treatment of patients with microsatellite instability-high (MSI-H) or mismatch repair-deficient (dMMR) unresectable or metastatic colorectal cancer. Eligible participants who meet the inclusion and exclusion criteria will provide written informed consent and receive QL1706 at 5.0 mg/kg and bevacizumab at 7.5 mg/kg on Day 1 of every 3-week cycle (Q3W), until disease progression or completion of 2 years of treatment. The primary endpoint of this study is objective response rate (ORR). Secondary endpoints include disease control rate (DCR), duration of response (DoR), progression-free survival (PFS), overall survival (OS), PFS and OS rates at 6, 12, and 24 months, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signs the informed consent form.
* Aged between 18 and 80 years (inclusive) at the time of consent; no gender restriction.
* Histologically confirmed unresectable locally advanced or metastatic colorectal cancer.
* At least one measurable target lesion according to RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* No prior immunotherapy for unresectable locally advanced or metastatic colorectal cancer.
* If previously treated with standard neoadjuvant or adjuvant therapy, the interval from the last dose to the first study treatment must be ≥ 6 months.
* Willing and able to provide tumor tissue and blood samples for MSI, RAS, BRAF, and PD-L1 testing.
* Estimated life expectancy of ≥ 12 months.
* Appropriate laboratory values must be met at screening.
* Female participants must be non-lactating, and have a negative pregnancy test result prior to enrollment.
* Participants of childbearing potential must agree to use effective contraception from the time of informed consent until at least 180 days after the last dose of study treatment.

Exclusion Criteria:

* Known history of severe allergic reactions to iparomlimab and tuvonralimab or bevacizumab.
* Active malignancy other than colorectal cancer within 5 years prior to first treatment.
* Large tumor lesions, especially those previously irradiated, with signs of bleeding.
* Imaging showing tumor invasion of major blood vessels (e.g., pulmonary artery or superior vena cava), including encasement or invasion of the vessel lumen.
* Brain metastases (asymptomatic or treated symptomatic brain metastases stable for >4 weeks allowed).
* Active autoimmune disease requiring systemic treatment.
* Active pulmonary diseases such as tuberculosis, radiation pneumonitis, drug-induced pneumonitis, or severe pulmonary dysfunction during screening.
* Requirement for long-term or high-dose NSAIDs (aspirin >325 mg) or anticoagulant therapy.
* History of severe gastrointestinal events within 6 months prior to first treatment.
* Severe intestinal obstruction symptoms or signs and unretrieved intestinal stents at screening.
* Cardiovascular or cerebrovascular diseases including but not limited to: NYHA class > II heart failure; unstable or severe angina; myocardial infarction or stroke within 6 months; atrial fibrillation or other arrhythmias requiring treatment; symptomatic superior vena cava syndrome; prolonged QT interval (male QT > 450 ms; female QTc > 470 ms); uncontrolled hypertension despite medication (SBP >140 mmHg and/or DBP >90 mmHg) or history of hypertensive crisis or encephalopathy.
* Known bleeding disorders or coagulopathies.
* Uncontrolled pleural, pericardial, or ascitic effusions requiring drainage.
* Active infection or unexplained fever >38.5°C at screening (cancer-related fever allowed).
* Use of systemic broad-spectrum antibiotics within 30 days prior to first treatment.
* Systemic corticosteroids (>10 mg prednisone equivalent daily) or immunosuppressants within 14 days prior to first treatment, or immunostimulants within 4 weeks.
* Major surgery, severe fractures, or therapeutic clinical trials within 4 weeks prior to first treatment; herbal treatment within 2 weeks.
* Ongoing adverse events from prior antitumor therapy greater than grade 1.
* HIV infection, other congenital or acquired immunodeficiencies, or history of organ or allogeneic bone marrow transplantation (except corneal transplantation).
* Positive hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) with HBV DNA >10⁴ copies/mL (~2000 IU/mL); or positive hepatitis C antibody with HCV RNA >10³ copies/mL; co-infection with HBV and HCV excluded.
* Vaccination with live or attenuated vaccines within 30 days prior to first treatment.
* Prior treatment with immune checkpoint inhibitors (e.g., anti-PD-1, anti-PD-L1, anti-CTLA-4, anti-OX-40, anti-CD137).
* Prior adjuvant targeted therapy against EGFR, VEGF, or VEGFR (e.g., bevacizumab, cetuximab, panitumumab, apatinib, regorafenib, anlotinib).
* Psychiatric disorders, epilepsy, dementia, or substance abuse that may affect compliance.
* Other conditions or lab abnormalities that may interfere with study participation or confound results as judged by investigators or sponsors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-06-27 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | approximately 6 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) according RESIST1.1 in total subjects

SECONDARY OUTCOMES:
DCR | approximately 12 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) and stable disease(SD) in total subjects
DOR | approximately 12 months after the last subject participating in
  The time from the date for first documented response of complete response (CR) or partial response (PR) to the date of first documented of disease progression or death, whichever occurs first.
PFS | approximately 12 months after the last subject participating in
  The time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first (per RECIST 1.1).
6/12/24 PFS rate | 6/12/24 months after the last subject participating in
  6/12/24 months survival rate based on PFS Kaplan-Meier curve
OS | approximately 12 months after the last subject participating in
  The time from the starting date of study drug to the date of death due to any cause.
6/12/24 OS rate | 6/12/24 months after the last subject participating in
  6/12/24 months survival rate based on OS Kaplan-Meier curve
Safety (adverse event) | Up to approximately 2 years
  The rates of adverse events based on NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China